CLINICAL TRIAL: NCT06817083
Title: Efficacy of Hook Technique Versus Traditional Methods for Single Hand Ventilation in Obese Patients a Randomized Controlled Trial
Brief Title: Comparison of Mask Ventilation in Obese Patients by Differents One Hand Techniques
Acronym: E&c / T&E
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Elhussein Mohammed Abdelkader, lecturer, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 964/9/24
Record Dates: First submitted 2025-01-06; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mask Ventilation
Keywords: mask ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group Hook technique (Active Comparator): novel method for single-hand ventilation that has shown promise in preliminary studies. This technique involves a unique hand positioning that aims to improve mask seal and ventilation efficacy, particularly in patients with challenging airway anatomy. In Hook Technique using the thumb and index finger to form a hook around the mask, creating a more secure and adjustable seal and utilizing the remaining fingers to apply consistent mandibular lift
  Interventions: Procedure: The Hook Technique
- Group E&c technique (Active Comparator): E-C clamp technique involves forming a "C" with the thumb and index finger around the mask while the remaining fingers form an "E" to lift the mandible. This technique aims to provide a good seal while opening the airway.
  Interventions: Procedure: E-C Clamp Technique
- Group T&E (Active Comparator): T-E technique is a variation where the thumb and index finger form a "T" over the mask while the other fingers provide chin lift and jaw thrust. This method is designed to optimize airway patency and mask seal.
  While these techniques are widely taught and practiced, they often fall short in obese patients due to the difficulty in maintaining an adequate seal and achieving sufficient ventilation pressures. Complications such as hypoxemia and gastric insufflation are more common in this population
  Interventions: Procedure: T-E Technique

INTERVENTIONS:
Procedure: E-C Clamp Technique — The E-C clamp technique involves forming a "C" with the thumb and index finger around the mask while the remaining fingers form an "E" to lift the mandible. This technique aims to provide a good seal while opening the airway.
  Arms: Group E&c technique
Procedure: T-E Technique — The T-E technique is a variation where the thumb and index finger form a "T" over the mask while the other fingers provide chin lift and jaw thrust.
  This method is designed to optimize airway patency and mask seal. While these techniques are widely taught and practiced, they often fall short in obese patients due to the difficulty in maintaining an adequate seal and achieving sufficient ventilation pressures. Complications such as hypoxemia and gastric insufflation are more common in this population.
  Arms: Group T&E
Procedure: The Hook Technique — e is a novel method for single-hand ventilation that has shown promise in preliminary studies. This technique involves a unique hand positioning that aims to improve mask seal and ventilation efficacy, particularly in patients with challenging airway anatomy. In Hook Technique using the thumb and index finger to form a hook around the mask, creating a more secure and adjustable seal and utilizing the remaining fingers to apply consistent mandibular lift, enhancing airway patency.
  Arms: Group Hook technique

SUMMARY:
The goal of this controled clinical trial study to know if hook tecnique method is better than other traditional one hand ventilation methods in acheiving effective ventilation in obese patients .

The main questions it aims to answer [are]:

Primary Outcome Measures

1. Success Rate of Ventilation:

   Definition: The primary measure of success will be defined as achieving effective ventilation within a set timeframe. Effective ventilation is indicated by:
   1. Visible and adequate chest rise and fall.
   2. chest expansion by ultra-sounded guided diaphragmatic excursion at certain time 30, 60, 90, 120 second.
   3. End tidal Co2 in Capnography at certain time 30, 60, 90, 120 second.
   4. Oxygen saturation (SpO2) levels reaching ≥ 95% within 2 minutes of applying the ventilation technique.
   5. Exhaled Tidal Volume at certain time 30, 60, 90, 120 second.
   6. Peak Inspiratory Pressure (PIP).

      Measurement:

      • Chest Rise and Fall: This will be visually assessed by an independent observer.

      evaluation the techniques based on the chest expansion score from 1 to 4. To evaluate Chest Rising in the studied patients, by visual method, patients were categorized into four groups: the amount of chest rising in group one was between 0 and 25% (score 1), 25-50% in group two (score 2), 50-75% in group three (score 3) and 75-100% in group four (score 4). Patients in group one and two considered to have unsuccessful ventilation due to lack in chest rise, and in groups three and four, the ventilation was considered successful • Ultra-sounded guided diaphragmatic excursion: It will be considered successful ventilation if Diaphragmatic excursion more than 2 cm and will be considered ventilation failure if less than 2 cm • Oxygen Saturation: SpO2 levels will be continuously monitored using a pulse oximeter, with readings recorded at baseline (before ventilation) and at regular intervals (every 15 seconds) until effective ventilation is achieved or the 2-minute mark is reached.

      • Measurement of Exhaled Tidal Volume: Determine if the Hook Technique provides superior tidal volume (mL/kg of predicted body weight) compared to the E-C and T-E techniques within the first 2 minutes of ventilation and will be consider successful ventilation if exhaled tidal volume more than 6 ml per kg and failure if less than 6 ml per kg

      • Peak Inspiratory Pressure (PIP): Compare the peak inspiratory pressures generated during ventilation with each technique and will be consider failure of ventilation if more than 30 Lower PIP for a given tidal volume indicates more efficient ventilation, which is particularly important in obese patients who often require higher pressures due to increased airway resistance Secondary Outcome Measures
      1. Time to Achieve Effective Ventilation:

         Definition: The time taken from the initiation of the ventilation technique to the point at which effective ventilation is confirmed.

         Measurement:

         • The stopwatch will start as soon as the anesthesiologist initiates the ventilation technique.

         • The time will be stopped when the criteria for effective ventilation (chest rise and fall, SpO2 ≥ 95%) are met.

         • This measure provides an indication of the efficiency of each technique in rapidly achieving effective ventilation.
      2. Rate of Ventilation Attempts:

         Definition: The number of attempts needed to achieve effective ventilation.

         Measurement:

         Each attempt is defined as a discrete application of the ventilation technique. Multiple attempts within the 2-minute timeframe will be recorded and analyzed. The number of attempts required to achieve successful ventilation will be compared across the three techniques to assess reliability and ease of achieving effective ventilation.
      3. Incidence of Ventilation Failure:

         Definition: Failure to achieve effective ventilation within the 2-minute timeframe.

         Measurement:

         Any cases where effective ventilation is not achieved within 2 minutes will be documented.

         The reasons for failure (e.g., difficulty in mask seal, inadequate chest rise) will be recorded and analyzed to understand the limitations of each technique.
      4. Complications:

      Document any airway trauma, hypoxem

DETAILED DESCRIPTION:
Study Methods

* Population of study: These prospective randomized controlled clinical trials will be conducted at Aswan University hospital on 375 obese patients:
* Study location: This is a prospective study that will be conducted at Aswan University Hospital. Fit Patients who will undergo surgeries with BMI >30 Age: between 18 and 60. Both genders. ASA I/II patients.
* Exclusion criteria:

Morbid obese patients with BMI > 40 Having facial anomalies. Patients with pre-existing diaphragmatic or respiratory disorders ASA III/IV.

- Methodology in details: A computer-generated randomization list will be used to randomize consented study participants on a 1:1:1 ratio to compare hook method versus E/C versus T/E technique.

The patients will be randomly assigned to 3 groups

* Group 1 hook method: Providers will be trained and standardized in the new hook technique for single-hand ventilation
* Group 2 (E/C): Providers will use the thenar eminence-chin lift technique
* Group 3 (T/E): Providers will use the thenar eminence-encircling technique

Preoperative:

After taking consent from the patients included in the study, all patients will receive pre-anesthesia airway evaluation before entering the operation room, and their interincisor distance, thyromental distance and Mallampati classification will be measured and recorded. Each patient will be asked to fast for at least 8 h and will be given no premedicationnoninvasive blood pressure, pulse oximetry (SpO2), end-tidal CO2 estimation (PETCO2), anesthetic agent analyzer will be attached to all patients.

Intraoperative:

After 3 min of preoxygenation, general anesthesia will be induced using 1-2 μg/kg fentanyl, 2-3 mg/kg propofol, and 0.6-1.2 mg/ kg rocuronium followed by different desirable face mask-ventilation after full relaxation with a mixture of 100% oxygen and 2% sevoflurane and ventilation parameters will be setted up, volume control ventilation mode, tidal volume 8ml/kg ideal body weight, RR 12. PEEP 5, fio2 100 %. Antisialogogues will be used before instrumentation of airway (atropine 0.5-1 mg). Oral airway will be inserted according to measurement from angle of the mouth to angle of the mandible to facilitate the ventilation and make it symmetrical.

Technique:

Two commonly used traditional methods for single-hand ventilation include:

1. E-C Clamp Technique: The E-C clamp technique involves forming a "C" with the thumb and index finger around the mask while the remaining fingers form an "E" to lift the mandible. This technique aims to provide a good seal while opening the airway.
2. T-E Technique: The T-E technique is a variation where the thumb and index finger form a "T" over the mask while the other fingers provide chin lift and jaw thrust.

   This method is designed to optimize airway patency and mask seal. While these techniques are widely taught and practiced, they often fall short in obese patients due to the difficulty in maintaining an adequate seal and achieving sufficient ventilation pressures. Complications such as hypoxemia and gastric insufflation are more common in this population.
3. The Hook Technique is a novel method for single-hand ventilation that has shown promise in preliminary studies. This technique involves a unique hand positioning that aims to improve mask seal and ventilation efficacy, particularly in patients with challenging airway anatomy. In Hook Technique using the thumb and index finger to form a hook around the mask, creating a more secure and adjustable seal and utilizing the remaining fingers to apply consistent mandibular lift, enhancing airway patency.

   * Does the research involve? Human participants Biological samples/Tissues Identifiable private data/Information
   * Type of consent of study participants:

Written consent No consent needed (Please justify) Oral consen

* Potential risks:

  1. Hypoventilation
  2. Desaturation
  3. Hypercarbia

     Confidentiality of data:

     Ensure patient privacy, confidentiality of data throughout the study and Informed consent: Ensure participants fully understand the study and provide informed consent before participation. 9. Study outcomes

     The following outcomes will be recorded:

     Primary Outcome Measures 1. Success Rate of Ventilation: Definition: The primary measure of success will be defined as achieving effective ventilation within a set timeframe. Effective ventilation is indicated by:
     1. Visible and adequate chest rise and fall.
     2. chest expansion by ultra-sounded guided diaphragmatic excursion at certain time 30, 60, 90, 120 second.
     3. End tidal Co2 in Capnography at certain time 30, 60, 90, 120 second. prior to surgery. On arrival at the operating room (OR), five-lead ECG, d) Oxygen saturation (SpO2) levels reaching ≥ 95% within 2 minutes of applying the ventilation technique.

     e) Exhaled Tidal Volume at certain time 30, 60, 90, 120 second. f) Peak Inspiratory Pressure (PIP).

     Measurement:

     • Chest Rise and Fall: This will be visually assessed by an independent observer.

     evaluation the techniques based on the chest expansion score from 1 to 4. To evaluate Chest Rising in the studied patients, by visual method, patients were categorized into four groups: the amount of chest rising in group one was between 0 and 25% (score 1), 25-50% in group two (score 2), 50-75% in group three (score 3) and 75-100% in group four (score 4). Patients in group one and two considered to have unsuccessful ventilation due to lack in chest rise, and in groups three and four, the ventilation was considered successful • Ultra-sounded guided diaphragmatic excursion: It will be considered successful ventilation if Diaphragmatic excursion more than 2 cm and will be considered ventilation failure if less than 2 cm Technique of Diaphragmatic Assessment

     a) Equipment: using ultrasound machine (Mindray DP 2200plus). use a low -frequency convex ultrasound probe (6-15 MHz) for diaphragmatic imaging. connect the probe to ultrasound machine with appropriate software for image acquisition and analysis. b) Procedure: position the patient in semi-recumbent or supine position. Apply ultrasound Gel to the skin overlying the diaphragm in the subcostal area. place the ultrasound probe in the subcostal region to obtain the longitudinal view of the diaphragm. Adjust the ultrasound settings for optimal image quality, including gain, depth, and focus. Record both B-mode and M-mode images during face mask ventilation. Record real-time images during various respiratory phases. Measure excursion as the difference in diaphragmatic position between inspiration and expiration.
     * Oxygen Saturation: SpO2 levels will be continuously monitored using a pulse oximeter, with readings recorded at baseline (before ventilation) and at regular intervals (every 15 seconds) until effective ventilation is achieved or the 2-minute mark is reached.
     * Measurement of Exhaled Tidal Volume: Determine if the Hook Technique provides superior tidal volume (mL/kg of predicted body weight) compared to the E-C and T-E techniques within the first 2 minutes of ventilation and will be consider successful ventilation if exhaled tidal volume more than 6 ml per kg and failure if less than 6 ml per kg
     * Peak Inspiratory Pressure (PIP): Compare the peak inspiratory pressures generated during ventilation with each technique and will be consider failure of ventilation if more than 30 Lower PIP for a given tidal volume indicates more efficient ventilation, which is particularly important in obese patients who often require higher pressures due to increased airway resistance Secondary Outcome Measures

  <!-- -->

  1. Time to Achieve Effective Ventilation:

     Definition: The time taken from the initiation of the ventilation technique to the point at which effective ventilation is confirmed.

     Measurement:

     • The stopwatch will start as soon as the anesthesiologist initiates the ventilation technique.

     • The time will be stopped when the criteria for effective ventilation (chest rise and fall, SpO2 ≥ 95%) are met.

     • This measure provides an indication of the efficiency of each technique in rapidly achieving effective ventilation.
  2. Rate of Ventilation Attempts:

     Definition: The number of attempts needed to achieve effective ventilation.

     Measurement:

     Each attempt is defined as a discrete application of the ventilation technique. Multiple attempts within the 2-minute timeframe will be recorded and analyzed. The number of attempts required to achieve successful ventilation will be compared across the three techniques to assess reliability and ease of achieving effective ventilation.
  3. Incidence of Ventilation Failure:

     Definition: Failure to achieve effective ventilation within the 2-minute timeframe.

     Measurement:

     Any cases where effective ventilation is not achieved within 2 minutes will be documented.

     The reasons for failure (e.g., difficulty in mask seal, inadequate chest rise) will be recorded and analyzed to understand the limitations of each technique.
  4. Complications:

     Document any airway trauma, hypoxemia episodes (Defined as SpO2 dropping below 90% at any time during the ventilation attempts. The frequency and duration of hypoxemia episodes will be recorded.), or other adverse events. Incidents of trauma such as lip lacerations, dental injury, or soft tissue damage will be documented. The severity and type of airway trauma will be recorded and compared among the three techniques.
  5. Ease of use:

     Assessed through a standardized provider questionnaire rating comfort and ease on a Likert scale and the provider will be asked to rate the used technique of mask ventilation from easy to neutral to fatigue on using 10.Sample size Primary Outcome Measure: Success Rate of Ventilation Definition: Achieving effective chest rise and SpO2 ≥ 95% within 2 minutes of initiating ventilation. Primary Comparison: Success rates of the hook technique versus E/C and T/E techniques.

     Assumptions for Sample Size Calculation:

     Baseline Success Rate (E/C and T/E Techniques): Based on previous studies and clinical experience, assume a success rate of approximately 70% for traditional techniques in obese patients. Expected Success Rate (Hook Technique): Hypothesized to be higher, for instance, around 85%. Significance Level (α): 0.05 (two-sided) Power (1 - β): 0.80 (80% power) Effect Size: The difference in success rates (15%). Total Sample Size: 375 patients, approximately 125 patients per group (Hook, E/C, T/E).Study Blinding 1. Blinding of Outcome Assessors:

     • Outcome assessors and data analysts will be blinded to the used technique and the provider will be blinded to effective ventilation parameters to reduce bias in the evaluation of outcomes.

     • Blinded assessors will perform data collection related to primary and secondary outcome measures, such as chest rising, diaphragmatic excursion, exhaled tidal volume, PIP, SpO₂ levels, and provider feedback. 2. Blinding of Participants and Providers:
     * Full blinding of participants and providers is not feasible due to the nature of the intervention.

     However, efforts will be made to minimize bias by standardizing procedures and training.
     * Providers will be trained to perform all three techniques to reduce performance bias.

       11. Statistical analysis Data analysis will be conducted using SPSS software version 22. We will collect and analyze demographic data, reporting success rates as frequencies and mean ± standard deviation.

     Primary Analysis:

     We will compare the success rates using chi-square tests.

     Secondary Analysis:

     We will compare time to effective ventilation using ANOVA or Kruskal-Wallis tests.

     We will analyze ease of use ratings and complication rates using appropriate statistical tests.

     Multivariate Analysis:

     We will djust for potential confounders such as age, sex, and BMI category.

     Ethical Considerations:

     Informed Consent: All participants will provide written informed consent. Ethical Approval: The study will be approved by the institutional review board (IRB).

     Safety Monitoring: A data and safety monitoring board (DSMB) will oversee the trial.

  12. Source of funding: Non. 13.Time plan:
* When to start? July 2024
* When expected to finish? March 202514.References:

Balafar M, Pouraghaei M, Paknezhad SP, Abad SN, Soleimanpour H. Evaluation the quality of bag-mask ventilation by E/C, T/E and hook technique (a new proposed technique). BMC anesthesiology. 2023 Nov 23;23(1):384. Bengü GA, Küçükosman G, Pişkin Ö, Okyay RD, Ayoğlu H. Difficult Mask Ventilation in Obese Patients: New Predictive Tests?. Haseki Tip Bulteni. (2019) Mar 1;57(1):15.Bülent Ecevit University Faculty of Medicine, Department of Anesthesiology and Reanimation, Zonguldak, Turkey Bharadwaj MS, Sharma M, Purohit S, Joseph A. Comparison of the effectiveness of two-handed mask ventilation techniques (CE versus VE) in obese patients requiring general anesthesia in an Indian population. Anesthesia Essays and Researches. (2022)Jan 1;16(1):167-71. Cheeseman JF, Webster CS, Pawley MD, Francis MA, Warman GR, Merry AF. Use of a new task-relevant test to assess the effects of shift work and drug labelling formats on anesthesia trainees' drug recognition and confirmation. Canadian Journal of Anesthesia/Journal canadien d'anesthésie. (2011) ;1(58):38-47. Hagberg, C. A., & Artime, C. A. (2014). Airway Management in the Adult. In: Hagberg and Benumof's Airway Management, 3rd Edition. Elsevier. Lafferty, K. A., & Jones, D. P. (2019). Innovative Airway Management Techniques: Initial Clinical Outcomes. Journal of Clinical Anesthesia, 58, 50-57. Soleimanpour M, Rahmani F, Bagi HR, Ala A, Mahmoodpoor A, Hassani F, Sharifi SM, Esfanjani RM, Soleimanpour H. Comparison of three techniques on facility of bag-mask ventilation: Thenar eminence, EO and EC. Anesthesiology and pain medicine. (2018) Aug;8(4).Anesth Pain Med. 2018 Aug; 8(4): e74226. Published online 2018 Aug 11. doi: 10.5812/aapm.74226

ELIGIBILITY:
Inclusion Criteria:

* bmi > 30

Exclusion Criteria:

* bmi>40

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Single-Hand Ventilation Using the Hook Technique Versus the E/C and T/E Techniques in Obese Patients | 9 Months
  The proportion of successful single-hand ventilations achieved using the hook technique compared to the E/C (thenar eminence-chin lift) and T/E (thenar eminence-encircling) techniques in obese patients.

SECONDARY OUTCOMES:
Time to Achieve Effective Ventilation Using the Hook Technique Versus E/C and T/E Techniques in Obese Patients | 9 Months
  The time (in seconds) required to achieve effective ventilation using the hook technique compared to the E/C and T/E techniques.
Number of Attempts Needed to Achieve Effective Ventilation Using the Hook Technique Versus E/C and T/E Techniques | 9 Months
  The number of attempts required to achieve effective ventilation using the hook technique compared to the E/C and T/E techniques.
Ease of use of the Hook Technique Compared to E/C and T/E Techniques as Rated by Anesthesiologists | 9 Months
  The ease of use of the hook technique compared to the E/C and T/E techniques, as rated by anesthesiologists on a Likert scale (1-5).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol